CLINICAL TRIAL: NCT06868316
Title: Optimizing Retention on Duty in Patients With Chronic Ankle Instability Using Auditory Biofeedback Gait Training: A Multisite Randomized Controlled Trial
Brief Title: Auditory Biofeedback Gait Training Individuals With Chronic Ankle Instability
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kentucky (Other)
Responsible Party: Principal Investigator, Danielle Torp, Assistant Professor, University of Kentucky
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 98018; CDMRP-OR230135 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2025-03-07; First posted 2025-03-10 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Ankle Sprains; Ankle Injuries and Disorders
MeSH Terms: conditions — Ankle Injuries; Disease | interventions — Walking; Running

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Active Comparator): Control group will wear the Loadsol Pros in-shoe insoles, with the auditory biofeedback function disabled
  Interventions: Other: Walking; Other: Rucking; Other: Running
- auditory biofeedback (AudFB) gait training (Experimental): AudFB group will wear the Loadsol Pros in-shoe insoles with the audible noise emitted from the iOS device
  Interventions: Other: Walking; Other: Rucking; Other: Running

INTERVENTIONS:
Other: Walking — Weeks 1-2, Sessions 1-4: The first condition will be walking with the speed self-selected based on "a comfortable pace to walk for exercise" as determined during the Baseline testing session. This speed will be held constant for the 10-minute walking portion prior to each condition but will be progressed for the remaining walking condition sessions (Sessions 2-4). The minimum speed will be limited to 1 mph.
Other: Rucking — Weeks 3-4, Session 5-8: The second condition will require participants to wear a standard rucksack equal to 20% of their body weight (minimum ruck weight: 15 pounds, maximum ruck weight: 45 pounds). The initial speed used during this condition will be self-selected based on "a comfortable pace to walk for exercise carrying this weight" as determined during the Baseline testing session.
Other: Running — Weeks 5-6, Sessions 9-12: The final condition is running. The self-selected running pace will be chosen as a pace that the participant can "sustain for a leisure run for 20 minutes," as determined at the Baseline testing session. Participants will only run for the 15-minute condition period.

SUMMARY:
The goal of this randomized clinical controlled trial is examine the effects of gait training with auditory biofeedback (AudFB) on gait biomechanics, clinical measures of ankle joint health, and patient-centered outcomes. The following specific aims will achieve this objective:

* Specific Aim 1: Determine if a 6-week gait training with AudFB intervention improves lower extremity biomechanics compared to a Control condition in participants with CAI.
* Specific Aim 2: Determine if a 6-week gait training with AudFB reduces talar cartilage deformation compared to a Control condition in participants with CAI.
* Specific Aim 3: Determine if a 6-week gait training with AudFB reduces episodes of ankle giving-way and reduces self-perceived severity of symptoms relative to a Control condition in participants with CAI.

Participants will:

* Complete 12 intervention sessions over a 6-week period of walking, ruck marching, and runninig.
* Complete testing sessions before and after the intervention, then after 6 and 12-months following the intervention.

DETAILED DESCRIPTION:
Background: Ankle injuries account for the highest musculoskeletal injuries among conventional and special warfare combatants. In the civilian population, 40% of lateral ankle sprain patients will develop chronic ankle instability (CAI). If the same frequency is true in military settings, then up to 36,800 service members develop CAI annually. CAI contributes to the total number of medically non-available service members, creates a substantial economic burden, impacts the quality of duty-relevant task performance, and generates a large population of service members who require long-term care after retirement. There are no evidence-based gait training interventions for patients with CAI despite abnormal biomechanical patterns leading to recurring injuries linked to ankle osteoarthritis (OA) development. Overall, the current rehabilitation strategies are insufficient for preventing complications following an ankle sprain.

Hypothesis/Objectives: The overall objective of this study is to examine the effects of gait training with auditory feedback (AudFB) on gait biomechanics, ankle joint health, and patient-centered outcomes. Our central hypothesis is that a 6-week (12 sessions) gait training program with AudFB will lead to short and long-term improvements in walking, rucking, and running biomechanics, talar cartilage deformation patterns, giving way episodes and severity of symptoms.

Specific Aims:

Aim 1: Determine if a 6-week gait training with AudFB improves lower extremity biomechanics compared to a Control condition in participants with CAI.

Aim 2: Determine if a 6-week gait training with AudFB reduces talar cartilage deformation compared to a Control condition in participants with CAI.

Aim 3: Determine if a 6-week gait training with AudFB reduces ankle giving-way episodes and severity of CAI symptoms relative to a Control condition in participants with CAI.

Study Design: Specific Aims 1-3 will be addressed using a single-blinded, multi-site randomized controlled trial design with data collected at the University of Kentucky (UK) and University of North Carolina at Charlotte (UNC Charlotte) (Figure 3). Patients with CAI will be randomized to the AudFB or Control group at a 1:1 allocation ratio (n=100; 50 UK and 50 UNC Charlotte). Participants will report to the UK Sports Medicine Research Institute or the UNC Charlotte Biodynamics Research Laboratory to complete outcomes for Specific Aims 1-3 at Baseline, Post-Intervention, and 6- and 12-Month Post-Intervention sessions, which will record: 1) lower extremity biomechanics during walking, rucking, and running, 2) talar articular cartilage deformation via ultrasonography, and 3) ankle giving way and patient-reported outcomes of CAI symptom severity. The AudFB group and Control group will complete 12 sessions of supervised gait training over 6 weeks and follow the same condition-based progression design. Each session will last roughly 25 minutes and begin with 10 minutes of walking followed by 15 minutes of the designated condition for that session (walking, rucking, or running). The AudFB group will receive real-time biofeedback derived from plantar forces of the lateral foot. The control group will be instructed to walk comfortably. Both groups will wear standard neutral athletic shoes and wireless in-shoe force insoles during every intervention session for standardization of testing procedures.

Impact and Military Benefit: The Investigators expect participants with CAI in the AudFB group will exhibit improvements in patient-centered outcomes and subsequent clinician-centered outcomes regarding biomechanics and ankle joint health. These findings will signal that our novel AudFB gait training protocol is critical to short- and long-term quality of life in patients with CAI. This study will provide a short-term impact by providing clinicians with an easily accessible and feasible tool to implement gait training to optimize return to duty in service members with CAI history. The long-term impact of this study will be related to the expansion of the rehabilitation paradigm by providing an evidence-based gait training protocol that has the potential to mitigate the early onset of ankle OA.

ELIGIBILITY:
Inclusion Criteria:

* Physically active adults (defined as participants reporting a score of =4 on the National Aeronautics and Space Administration (NASA) Activity Instrument and indicating they can run for at least 20 consecutive minutes)
* History of ankle sprain
* 2 episodes of "giving way" in the past 6-months
* must answer "yes" to =5 questions on the Ankle Instability Instrument (AII) and =11 on the Identification of Functional Ankle Instability (IdFAI)

Exclusion Criteria:

* an ankle sprain in the previous four weeks or lower extremity neuromusculoskeletal injury other than to the ankle in the last 12 months
* history of surgery in the lower extremity
* fracture to the lower extremity in the past 12 months or a fracture that required open-reduction internal fixation
* history of neurological disease, vestibular or visual disturbance or any other pathology that would impair sensorimotor performance or gait
* current participation in a formal ankle joint rehabilitation program
* a concussion in the last 12 months
* report a cardiovascular, metabolic, or renal disease, or signs and symptoms that suggest such condition or have been told by a medical provider not to engage in vigorous physical activity (such as running).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-05-27 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Change in lower extremity biomechanics - peak pressure | baseline, immediately following the intervention, 6 months post intervention, and 12 months post intervention
  The assessment will consist of a 45-minute treadmill loading protocol with 15 minutes of each: walking, running, and ruck marching.
Change in lower extremity biomechanics - maximum force | baseline, immediately following the intervention, 6 months post intervention, and 12 months post intervention
  The assessment will consist of a 45-minute treadmill loading protocol with 15 minutes of each: walking, running, and ruck marching.
Change in lower extremity biomechanics - pressure-time integral | baseline, immediately following the intervention, 6 months post intervention, and 12 months post intervention
  The assessment will consist of a 45-minute treadmill loading protocol with 15 minutes of each: walking, running, and ruck marching.
Change in lower extremity biomechanics - force-time integral | baseline, immediately following the intervention, 6 months post intervention, and 12 months post intervention
  The assessment will consist of a 45-minute treadmill loading protocol with 15 minutes of each: walking, running, and ruck marching.
Change in Talar cartilage deformation | baseline, immediately following the intervention, 6 months post intervention, and 12 months post intervention
  Participants will be placed in a long-sitting position on a table for 30 minutes to limit the influence of the preceding activity on resting thickness volume. After the offloading period, participants will be positioned with their back flat against a wall, the test limb with the knee flexed at 90°, and their foot flat on a table. A 12-MHz linear ultrasound probe will be positioned transversely between the medial and lateral malleoli and adjusted until the talar cartilage appears to be maximum reflected. Images will be taken and averaged to assess structural and functional components of ankle joint health.
Change in self perceived ankle instability | Baseline, 6-Month Post-Intervention, and 12-Month Post-Intervention
  Ankle instability will be measured by the Cumberland Ankle Instability Tool (CAIT). This tool is designed to capture the severity of CAI through the 9-item scale focusing on the degree of difficulty in performing various physical activities due to the ankle. Scores range from 0 to 30, with a higher score indicative of higher stability
Change in self perceived foot and ankle disability | Baseline, 6-Month Post-Intervention, and 12-Month Post-Intervention
  The Foot and Ankle Disability Index (FADI) is a region-specific patient-reported outcome designed to assess functional limitations during activities of daily living and sports-related activities in participants with foot and ankle pathologies

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Kentucky, Lexington, Kentucky
  - University of North Carolina at Charlotte, Charlotte, North Carolina

IPD SHARING:
Plan to Share IPD: No